CLINICAL TRIAL: NCT05244057
Title: A Phase II of Randomized, Double-blind, Placebo-controlled, Multi-center Study of Hepalatide for Injection Combined With Pegylated Interferon and TAF as Finite Treatment in Chronic Hepatitis B Patients
Brief Title: A Study of Hepalatide Combined With TAF and PEG-IFN as Finite Treatment of Chronic Hepatitis B Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai HEP Pharmaceutical Co., Ltd. (Industry)
Collaborators: Shanghai Tong Ren Hospital (Other); Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: L47-HB-FIN-1(New Finite)
Record Dates: First submitted 2022-02-03; First posted 2022-02-17 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2023-12

CONDITIONS: Chronic Hepatitis B
Keywords: hepalatide, Hepatitis B，finite treatment,
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hepalatide + TAF + PEG-IFN (Experimental): Patients will receive 6.3mg Hepalatide +25mg Tenofovir alafenamide+ 90ug Pegylated Interferon for 48 weeks with a further follow-up period of 24 weeks.
  Interventions: Drug: Hepalatide; Drug: Tenofovir Alafenamide Tablets; Drug: Pegylated Interferon alfa 2a
- Placebo+ TAF + PEG-IFN (Placebo Comparator): Patients will receive Placebo +25mg Tenofovir alafenamide + 90ug Pegylated Interferon for 48 weeks with a further follow-up period of 24 weeks.
  Interventions: Drug: Placebo of Hepalatide; Drug: Tenofovir Alafenamide Tablets; Drug: Pegylated Interferon alfa 2a

INTERVENTIONS:
Drug: Hepalatide — 6.3mg, s.c., qd for 48 weeks
  Other Names: L47
  Arms: Hepalatide + TAF + PEG-IFN
Drug: Placebo of Hepalatide — s.c., qd for 48 weeks
  Other Names: Placebo
  Arms: Placebo+ TAF + PEG-IFN
Drug: Tenofovir Alafenamide Tablets — 25mg, p.o., qd for 48 weeks
  Other Names: Vemlidy
Drug: Pegylated Interferon alfa 2a — 90ug, s.c., qw for 48 weeks
  Other Names: Pegasys

SUMMARY:
The study is designed to assess efficacy of a finitie treatment in Chronic Hepatitis B patients who had stable treatment of NAs for ≧ 2 years， which is compared hepalatide in combination with Pegylated Interferon + TAF with Pegylated Interferon +TAF. Subjects will be randomly assigned to the hepalatide or placebo groups , 15 subjects in each group . Subjects will receive hepalatide+Pegylated Interferon +TAF treatment for 48 weeks or placebo +PegylatedInterferon +TAF treatment for 48 weeks , Then, stopping hepalatide and Pegylate Interferon treatments and followed with further 8 weeks follow-up.

DETAILED DESCRIPTION:
Hepalatide is a liver-targeted antiviral therapeutic for subcutaneous injection designed to treat chronic hepatitis B virus (HBV) infection. The aim of this study is to assess efficacy of a finitie treantment , that combination regimen of hepalatide+half dose Pegylated interferon + TAF , as measured by the primary efficacy endpoint. This study will be conducted in 3 periods: Screening Period (4weeks), Treatment Period (48 weeks) and Follow-up (FU) Period (8 weeks). Safety assessments will include adverse events (AEs), serious AEs, clinical safety laboratory tests, electrocardiograms (ECGs), vital signs, ophthalmologic examinations and physical examinations. Total duration of individual participation will be up to 60 weeks (including screening period).

ELIGIBILITY:
Inclusion Criteria:

* 1. HBsAg or/and HBV DNA Positive for at least 6 months

  2. HBeAg negative

  3. Received NAs stabilization therapy for at least 2 years

  4. ALT≤ 2×ULN

  5. HBV DNA< LLQD(lower limit of quantitative detection) in Screening

  6. Serum total bilirubin<2×ULN

  7. no childbirth plan within 2 years and agree to take effective contraceptive measures throughout the treatment period and within 3 months after the last dose, and that the woman is not pregnant or breastfeeding.

  8. have not participant in another clinical trial within 3 months before screening

  9. Subjects have good compliance with the protocol

  10. Subjects understood and agreed to sign the informed consent form.

Exclusion Criteria:

* 1. Contraindications of Peginterferon such as depressive disorder, epilepsy, autoimmune diseases, uncontrolled thyroid dysfunction, etc

  2. Subjects with cirrhosis, e.g., definite cirrhosis on imaging such as abdominal ultrasound and CT; liver biopsy with Metavir fibrosis score = 4; clinical diagnosis of cirrhosis by the investigator.

  3. Decompensated liver disease

  4. Child-Pugh score of B-C or over 6 points.

  5. Subjects with any of the following circumstances
* History of decompensated liver disease
* History of serious heart disease (including unstable or uncontrolled heart disease within 6 months)
* Uncontrolled seizures, severe psychiatric disorders, or a history of psychiatric disorders
* with history of organ transplantation
* with poorly controlled diabetes and hypertension
* with autoimmune diseases, immune-related extrahepatic manifestations, thyroid disease, malignant tumors, or in immunosuppressive therapy
* underlying diseases such as malignant tumor, severe infection, heart failure and chronic obstructive pulmonary disease and other serious diseases.
* with history of alcohol or drug abuse

  6. Creatinine clearance <60 mL/min.

  7. HAV, HCV, HDV, HEV or HIV co-infection

  8. Subjects who must be treated with Nucleosides (acids) other than TAF during treatment period

  9. Subjects who used interferon in the 6 months prior to the screening period

  10. Positive for anti-HBV Pre-S1 antibody.

  11. Hemocytopenia: White blood cells < 3 × 10^9 / L, neutrophil < 1.5 × 10^9 / L, platelet < 60 × 10^9 / L,

  12. Female subjects pregnancy test positive

  13. known to be allergic to the investigational drug or the underlying treatment drug

  14. Other laboratories or auxiliary examinations are obviously abnormal

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with negative conversion of HBsAg | 56 Weeks
  Proportion of subjects with negative conversion of HBsAg treatment at 8 weeks off treatment

SECONDARY OUTCOMES:
Number of subjects with virological relapse(VR) at 8 weeks off treatment | 56 Weeks
  VR: reappearance of HBV DNA > 2000 IU/ml from undetectable status
Number of subjects with clinical relapse(CR) at 8 weeks off treatment | 56 Weeks
  CR: the presence of VR with the elevation of alanine transaminase (ALT) more than two times upper limit of normal (ULN)
HBsAg is down from baseline at 8 weeks off treatment | 56 Weeks
  HBsAg is down from baseline log10
Number of subjects with Serological conversion of HBsAg | 56 Weeks
  Number of subjects with Serological conversion of HBsAg at 8 weeks off treatment
Change in liver stiffness at 8 weeks off treatment | 56 Weeks
  The findings of Liver stiffness measurement(LSM) of Fibroscan/FibroTouch at week 8 off treatment compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Qin Zhang, Principal Investigator — Shanghai Tong Ren Hospital
Locations (1):
- Shanghai Tong Ren Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No